CLINICAL TRIAL: NCT01098084
Title: A Phase II Study of Decitabine in Patients With Chronic Myelomonocytic Leukemia
Brief Title: Decitabine in Patients With Chronic Myelomonocytic Leukemia (CMML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Eric Solary, MD PhD, Unite INSERM 1009 Institut Gustave Roussy
Allocation: Not Applicable | Model: Single Group
Other Study IDs: GFM-DEC-LMMC-2007
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Myelomonocytic Leukemia
Keywords: Decitabine, chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine (Experimental)
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20mg/m2/day, one hour intravenous infusion, every day during 5 days

SUMMARY:
The aim of this study is to determine the therapeutic efficacy of Decitabine in patients with chronic myelomonocytic leukemia (CMML) diagnosis according to WHO criteria either untreated or previously treated with Hydrea or Etoposide (given orally), non intensive chemotherapy or intensive chemotherapy given more than 3 months before inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* CMML diagnosis according to WHO criteria
* Stable excess in blood monocytes,>1x10G/l and >10% of WBC
* Bone marrow blasts <20%
* Dysplasia of at least one lineage or clonality marker or blood monocytosis during more than 3 months w/o other explanation
* With:

  * if WBC < or= 12 000/mm3: IPSS high or intermediate 2
  * if WBC > 12 000/mm3: at least two of the following criteria: blast cells > 5% in the bone marrow, clonal cytogenetic abnormality other than t(5;12)(q33;p13), anemia (Hb < 100 g/l), thrombocytopenia (platelet count < 100G/l), splenomegaly > 5 cm below costal margin, extramedullary localization
* Either untreated or previously treated with
* Hydrea or Etoposide given orally
* non intensive chemotherapy
* intensive chemotherapy given more than 3 months before inclusion
* With performance status 0-2 on the ECOG scale
* With estimated life expectancy of at least 12 weeks
* With adequate organ function including the following:

  * Hepatic: total bilirubin < 1.5 times upper limit of normal (ULN), alanine transaminase (ALT) and aspartate transaminase (AST) < 3 times ULN
  * Renal: serum creatinine < 1.5 times ULN, creatinine clearance > 30 ml/min
* With informed consent
* Negative pregnancy and adequate contraception if relevant

Exclusion Criteria:

* Myeloproliferative/myelodysplastic syndrome other than CMML
* Acute blastic transformation of CMML with bone marrow blasts>20%
* Patients eligible for allogenic bone marrow transplantation with identified donor
* CMML with t(5;12) or PDGFbetaR rearrangement that could receive Imatinib
* Previous treatment with a hypomethylating agent
* Age < 18 years old
* Pregnancy or breastfeeding
* Performance status> 2 on the ECOG Scale
* Estimated life expectancy < 12 weeks
* Serious concomitant systemic disorder, including active bacterial, fungal or viral infection, that in the opinion of the investigator would compromise the safety of the patient and/or his/her ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine response of patients with CMML to 6 courses of Decitabine according to IWG 2006 criteria, adapted for CMML with WBC>12000/mm3

SECONDARY OUTCOMES:
Response duration
Time to progression to AML
Survival
Toxicity (hematological and non-hematological)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Solary, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Thorsten Braun, MD,PhD, Principal Investigator — Avicenne Hospital, 93 000 Bobigny; Ingrid Lafon, MD, Principal Investigator — CHU Le Bocage, Dijon
Locations (31):
- France (31):
  - CHR La Source orléans, Orléans, Orléans
  - CHU d'Amiens, Amiens
  - CH Angers, Angers
  - Hôpital Avignon, Avignon
  - Hopital de la Cote Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU Haut-Lévèque, Bordeaux
  - Hôpital Boulogne Sur Mer, Boulogne-sur-Mer
  - Hopital d'Instruction des Armées Percy, Clamart
  - CHU de, Clermont-Ferrand
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Hôpital Versailles, Le Chesnay
  - Centre Hospitalier du Mans, Le Mans
  - Institut Paoli Calmettes, Marseille
  - CHU de nantes, Nantes
  - Hôpital Archet1, Nice
  - CHU Caremeau, Nîmes
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - Hopital Hotel Dieu, Paris
  - Hoiptal St Louis, Paris
  - Hôpital Saint-Antoine., Paris
  - Centre Hospitalier Joffre, Perpignan
  - CHU de Reims, Reims
  - Centre Henri Becquerel, Rouen
  - Hematology Dpt, Hopital Purpan, Toulouse
  - CHU Bretoneau, Tours
  - Institut gustave Roussy, Villejuif
  - CHU de Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region

REFERENCES:
- [Derived] Itzykson R, Kosmider O, Renneville A, Gelsi-Boyer V, Meggendorfer M, Morabito M, Berthon C, Ades L, Fenaux P, Beyne-Rauzy O, Vey N, Braun T, Haferlach T, Dreyfus F, Cross NC, Preudhomme C, Bernard OA, Fontenay M, Vainchenker W, Schnittger S, Birnbaum D, Droin N, Solary E. Prognostic score including gene mutations in chronic myelomonocytic leukemia. J Clin Oncol. 2013 Jul 1;31(19):2428-36. doi: 10.1200/JCO.2012.47.3314. Epub 2013 May 20. PMID 23690417
- [Derived] Braun T, Itzykson R, Renneville A, de Renzis B, Dreyfus F, Laribi K, Bouabdallah K, Vey N, Toma A, Recher C, Royer B, Joly B, Vekhoff A, Lafon I, Sanhes L, Meurice G, Orear C, Preudhomme C, Gardin C, Ades L, Fontenay M, Fenaux P, Droin N, Solary E; Groupe Francophone des Myelodysplasies. Molecular predictors of response to decitabine in advanced chronic myelomonocytic leukemia: a phase 2 trial. Blood. 2011 Oct 6;118(14):3824-31. doi: 10.1182/blood-2011-05-352039. Epub 2011 Aug 9. PMID 21828134